CLINICAL TRIAL: NCT03475667
Title: Comparison of Radial and Femoral Artery Site Invasive Blood Pressure Measurement in Septic Patients on High Dose of Noradrenaline: A Prospective Observational Study
Brief Title: Comparison of Radial and Femoral Artery Site Invasive Blood Pressure Measurement in Septic Shock Patients
Status: Completed | Type: Observational
Sponsor: Sanjay Gandhi Postgraduate Institute of Medical Sciences (Other Government)
Responsible Party: Principal Investigator, Mohan Gurjar, Professor, Sanjay Gandhi Postgraduate Institute of Medical Sciences
Other Study IDs: 2018-27-DM-EXP
Record Dates: First submitted 2018-03-18; First posted 2018-03-23 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Septic Shock
Keywords: Septic Shock; hemodynamic monitoring; blood pressure determination
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Inaccurate monitoring of mean arterial pressure (MAP) could lead to improper treatment in the form of excessive fluid infusion or unnecessary vasopressor therapy; therefore, accurate hemodynamic monitoring is crucial in treatment of septic shock.

In critically ill septic patients treated with vasoactive drugs, many studies reported that radial arterial pressure monitoring significantly underestimates central arterial pressure. Insertion of a femoral line allowed a substantial reduction of the infusion rate of vasoactive drugs in these patients. These findings might imply that femoral placement of arterial lines is the gold standard for invasive arterial blood pressure monitoring in shock patient.

Our study aimed to determine the difference between radial (peripheral) and femoral (central) arterial pressures measured simultaneously in a group of critically ill patients receiving high dose noradrenaline therapy (≥ 0.1 mcg/kg/min).

DETAILED DESCRIPTION:
Invasive arterial blood pressure monitoring is common in critically ill patients admitted in intensive care units (ICUs). The most common indication for invasive arterial blood pressure monitoring is for continuous measurement in hemodynamically unstable patients on vasopressor therapies Invasive arterial blood pressure monitoring is a standard of care during shock management in the ICU. The Surviving Sepsis Campaign international consensus guidelines (2016) recommend maintaining a mean arterial pressure (MAP) of 65 mmHg or greater, as a goal of initial resuscitation, and to apply vasopressors, if required, to maintain MAP at this level. The radial artery is most commonly used, with the femoral artery being the second choice; both site accounting as 92% of all arterial cannulations.

Accuracy of invasive blood pressure monitoring is crucial in evaluating the cardiocirculatory system and adjusting vasopressor therapy for hemodynamic support. However, the best site for catheter insertion is controversial. Compared with arterial pressure waveforms measured in the central arteries (eg, aorta or femoral artery), those at the periphery (eg, radial artery) characteristically have steeper upstrokes, higher systolic peaks, a later appearing diastolic notch, more prominent diastolic waves and lower end-diastolic pressure. Yet, under normal physiological conditions, only a negligible decrement in MAP occurs. In critically ill patients during aberrant hemodynamic conditions like septic shock, gradients in MAP may develop from the central to the peripheral arterial site.

There are some available studies where simultaneous measurement of radial and femoral was done in different patient population. In all studies where patients of cardiopulmonary bypass were included showed that there was significant difference in MAP and SBP between femoral and radial invasive blood pressure measurements with femoral site IBP being greater than radial site. Similar difference in SBP and MAP was noted in reperfusion stage of liver transplant patients. The difference was also found in septic shock patients in MAP with vasopressor usage but one study did not find significant difference in invasive MAP and SBP.

Work plan methodology:

This is a prospective observational study to know the difference in blood pressure recordings of invasive arterial BP (radial versus femoral site) in patients of septic shock on high dose of noradrenaline therapy (≥0.1 mcg/kg/min) for at least 30 minutes. Participant will be included from ICU of department of critical care medicine. All adult critically ill patients with septic shock requiring noradrenaline infusion (≥0.1 mcg/kg/min) will be considered for inclusion in this study. Participant will be included if treating team considered to change the site of arterial invasive blood pressure monitoring from radial to femoral site (same side, left or right).

All three measurements: systolic blood pressure (SBP), diastolic blood pressure (DBP) and mean blood pressure (MAP) will be recorded three times, simultaneously on the monitor within 5 minutes of placement of femoral arterial catheter by freezing/taking snapshot of the monitor. Measurement will be recorded in supine position, with radial arterial line transducer at the level of 5th rib in mid-axillary line. Femoral line transducer will be placed at the same level as radial line transducer; the equality of the levels of both the transducers will be confirmed with the help of spirit level technique. Investigators will use 20 gauge arterial cannula for radial artery cannulation and 16 gauge single lumen catheters for femoral artery cannulation with all aseptic precautions. Participant with any change in noradrenaline dose requirement during study period (measurement of pressures) will be excluded from the analysis

Sample size and statistical analysis:

From the previous observational study considering minimum average difference of mean MAP of 2.8 mm of Hg, investigators calculated the sample size with power analysis by using version 2008 (PASS-8). A sample size of 44 achieves 90% power to detect a mean of paired differences of 2.8 with an estimated standard deviation of differences of 5.6 and with a significance level (alpha) of 0.05 using a two-sided paired t-test. In this study, investigators would also like to do the subgroup analysis in patients on very high dose of noradrenaline (≥0.3 mcg/kg/min). So, investigators will include 80 patients. Mean of three recordings each of SBP, DBP and MBP will be calculated and appropriate statistical methods will be applied

Intervention:

None

Duration of the study:

21 months

ELIGIBILITY:
Inclusion Criteria:

* All ICU patients who are ≥18 years with septic shock on high dose of noradrenaline (≥0.1 mcg/kg/min) for at least 30 minutes

Exclusion Criteria:

* Age <18 years
* Pregnancy
* Patient who cannot be made supine as per clinical condition
* Patients having abdominal compartment syndrome
* Known peripheral vascular disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients having septic shock on high dose of noradrenaline (≥0.1 mcg/kg/min) for at least 30 minutes.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2018-04-11 (Actual); Primary Completion 2020-01-10 (Actual); Study Completion 2020-01-10 (Actual)

PRIMARY OUTCOMES:
To compare radial and femoral arterial invasive blood pressure measurements in patients receiving high dose of noradrenaline (≥ 0.1 mcg/kg/min). | Within 5 minutes of placement of femoral artery catheter
  Comparison of radial and femoral artery site invasive blood pressure measurement in septic patients on high dose of noradrenaline

CONTACTS AND LOCATIONS:
Overall Officials: Mohan Gurjar, MD, PDCC, Principal Investigator — Sanjay Gandhi Postgraduate Institute of Medical Sciences (SGPGIMS)
Locations (1):
- Department of Critical Care Medicine, SGPGIMS, Lucknow, Uttar Pradesh, India

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Bhaskar B, Gurjar M, Mishra P, Azim A, Poddar B, Baronia AK. Arterial site selection for measurement of mean arterial pressure in septic shock patients on high-dose norepinephrine. Front Med (Lausanne). 2022 Dec 23;9:1019752. doi: 10.3389/fmed.2022.1019752. eCollection 2022. PMID 36619630